CLINICAL TRIAL: NCT06829082
Title: Clinical Effectiveness, Adherence, Clinical and Paraclinical Outcomes Associated With Tenofovir Alafenamide/Emtricitabine/Bictegravir (TAF/FTC/BIC) in Patients Diagnosed With Human Immunodeficiency Virus HIV) in Colombia: A Real-Life Study
Brief Title: Real-Life Outcomes of TAF/FTC/BIC in HIV Patients in Colombia
Status: Completed | Type: Observational
Sponsor: Servicios de Salud IPS Suramericana S.A.S (Other)
Responsible Party: Sponsor
Other Study IDs: SR-GL-003
Record Dates: First submitted 2025-02-03; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: HIV Treatment
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: BIKTARVY 50Mg-200Mg-25Mg Tablet — Antiretroviral therapy (ART) has advanced with the introduction of integrase strand transfer inhibitors (INSTIs), such as the fixed-dose combination of tenofovir alafenamide/emtricitabine/bictegravir (TAF/FTC/BIC), known as Biktarvy®. This regimen is preferred for its high genetic barrier to resistance, minimal drug interactions, and once-daily, single-tablet formulation, which enhances adherence and long-term treatment outcomes. While clinical trials have demonstrated its efficacy, real-world data specific to Colombia are lacking.

SUMMARY:
HIV remains a major global health issue, with 38 million people affected, and significant challenges in diagnosis and treatment due to stigma and socioeconomic factors. In Colombia, the epidemic is concentrated among men who have sex with men, with 165,405 people living with HIV and 14,670 new cases reported in 2023. Barriers to treatment access are exacerbated by social factors and Venezuelan migration. While integrase inhibitors like TAF/FTC/BIC have shown effectiveness, real-world data in Colombia is limited. This study evaluates adherence, effectiveness, and clinical outcomes of TAF/FTC/BIC in 169 patients within the EPS SURA program, contributing context-specific evidence.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older.
* Individuals with a confirmed HIV diagnosis.
* Individuals enrolled in EPS SURA during the study period.
* Patients receiving treatment with the TAF/FTC/BIC regimen.

Exclusion Criteria:

* Patients with a concurrent diagnosis of tuberculosis.
* Pregnant patients during the study period.
* Patients with virologic failure.
* Patients who started treatment with TAF/FTC/BIC but changed providers or discontinued treatment before completing six months of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the defined selection criteria within the established time frame for the search will be included.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Effectiveness: Virological Suppression | From enrollment to weeks 24 and 48
Effectiveness: CD4 T-Lymphocytes count | From enrollment to weeks 24 and 48
Security: Treatment-Related Adverse Events | From enrollment to weeks 24 and 48

SECONDARY OUTCOMES:
Security: Paraclinical Results: Hepatic and Renal Function, and Lipid Profile | From enrollment to weeks 24 and 48
  The lipid profile will be evaluated using HDL and LDL levels before the start of treatment and at 24 and 48 weeks of treatment.
Adherence to Treatment | From enrollment to week 48
  Adherence will be measured using pharmacy claims information with the Proportion of Days Covered (PDC). PDC calculates the proportion of days the patient has access to the medication over a specified period.
Security; Hepatic function | From enrollment to week 48
  Liver function will be evaluated by AST and ALT enzymes and total bilirubin levels before the start of treatment and at 24 and 48 weeks of treatment.
Security: Renal function | From enrollment to weeks 24 and 48
  Renal function will be assessed by serum creatinine levels before the start of treatment and at 24 and 48 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Servicios de Salud IPS Suramericana S.A.S., Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Following the results of the study, they will be analyzed and evaluated by the team designated for this purpose. When the final version of the study product has been obtained and the draft manuscript has been reviewed and approved by the authors, it will be submitted to the journal selected and agreed upon by the principal investigator, according to the impact classification of the publication. In addition, it will be presented at a previously selected scientific event (congresses, symposia, among others).
  Publications will comply with the guidelines of the International Committee of Medical Journal Editors (ICMJE). Likewise, all individuals who meet the authorship criteria defined by the ICMJE will be recognized as authors of the publications (http://www.icmje.org).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT06829082/Prot_SAP_000.pdf